CLINICAL TRIAL: NCT07253194
Title: Effect of Electroacupuncture on Postoperative Urinary Retention After Radical Surgery for Cervical Cancer： A Randomized Controlled Trial
Brief Title: Electroacupuncture on Postoperative Urinary Retention After Radical Surgery for Cervical Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lu Chao (Other)
Responsible Party: Sponsor-Investigator, Lu Chao, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2025-1315
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Urinary Retention (POUR)
Keywords: Postoperative urinary retention; POUR; Electroacupuncture; EA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The EA Group (Experimental): Participants will receive the EA intervention for two consecutive weeks.
  Interventions: Other: EA intervention
- The sham EA Group (Sham Comparator): Participants will receive the sham EA intervention for two consecutive weeks.
  Interventions: Other: Sham EA intervention

INTERVENTIONS:
Other: EA intervention — Participants will undergo EA treatment. Acupoint selection: Shenshu(BL23), Pangguanghu (BL28), Ciliao (BL32), Zhongliao (BL33), Huiyang (BL35), and Zhibian (BL54). Acupuncture needles (0.30 × 50 mm) will be vertically inserted into BL32, BL23, BL28, and BL35 at a depth of 40 ± 8 mm. The disposable acupuncture needle (0.45 × 75 mm) will be inserted into BL54 at a depth of 55 ± 10 mm, with the direction of insertion toward Shuidao (ST28). EA will be applied to the BL32 and BL54 points on both sides of the spine at a frequency of 2 Hz and a stimulation intensity of 2 ± 1.5 mA. Each treatment will last for 30 minutes, 5 days per week, for 2 weeks. Follow-up will be performed 2 weeks after the final treatment.
  Arms: The EA Group
Other: Sham EA intervention — Participants will receive sham EA treatment. Acupoint selection: consistent with the EA group. Sham acupuncture procedure: The disposable acupuncture needle (0.25 × 40 mm) will be used, and all acupoints will be shallowly penetrated into the skin using a vertical method, with a needle depth of 5 ± 2 mm. Sham EA application: EA electrodes will be attached identically to the EA group at a frequency of 2 Hz and a nominal intensity of 2 mA. However, no electrical current will be delivered via the EA device, as the connecting wires will undergo specialized modification. Each treatment session will also last 30 minutes, 5 days per week, for 2 weeks. The Follow-up will also be performed 2 weeks after the final treatment.
  Arms: The sham EA Group

SUMMARY:
This is a prospective, blinded, single-center, randomized controlled trial. Investigators will include 208 patients with postoperative urinary retention (POUR) after radical hysterectomy for cervical cancer who have a clear diagnosis and meet the screening criteria. Participants will be randomly divided into the electroacupuncture（EA）group and the sham EA group according to a 1:1 ratio. Each group consists of 104 patients, and all participants will be required to sign a written informed consent form. The TEAS group will be treated with EA based on conventional treatment, and the shamEA group will be treated with sham EA based on conventional treatment. The main outcomes will be to calculate the proportion of patients who successfully removed the urinary catheter, and the secondary indicators will include the change in post-void residual (PVR) volume of the bladder, assessment of urinary tract infection (UTI), and quality of life assessment according to the EORTC QLQ-C30 scale. Evaluation of participant-reported expectations, blinding, compliance, and safety will also be conducted. All analyses will be conducted in accordance with the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* ① 18 to 70 years old;
* ② Anticipated survival of at least 6 months;
* ③ Met the diagnostic criteria for POUR of cervical cancer, and the duration of POUR is less than 6 months;
* ④ No serious urinary system disease in the past, and no urinary retention before operation;
* ⑤ Karnofsky functional status score (KPS) ≥ 70 points;
* ⑥ Stable vital signs, no serious mental illness, capable of daily living, able to cooperate in completing all treatments and examinations;
* ⑦ Voluntarily participate and sign a written informed consent form.

Exclusion Criteria:

* ① Obstructive urinary retention, such as urethral stricture or stones induced urinary system diseases;
* ② Merge other serious systemic diseases, and advanced cachexia patients;
* ③ Patients who are intolerant to electrical stimulation therapy, such as those with pacemakers installed;
* ④ With psychiatric disorder or severe cognitive impairment;
* ⑤ Severe skin damage, infection, and ulceration at the treatment site;
* ⑥ Those who are participating in other acupuncture or drug clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The response rate of participants who will successfully remove the urinary catheter | week 0（baseline），and week 2 (after intervention)
  The participants in each group who will remove their urinary catheters after intervention, in proportion to the total number of patients in each group, multiplied by 100%. It can also be understood as the initial cure rate of POUR. The standard for patients to remove the urinary catheter is that the PVR volume is less than 100ml.

SECONDARY OUTCOMES:
The changes in PVR volume. | week 0 (baseline), week 2 (after intervention), and week 4 （follow-up）
  It will be measured by professional nurses, using a direct measurement method.
Assessment of UTI. | week 0 (baseline), week 2 (after intervention), and week 4 （follow-up）
  Urinalysis or urine culture will be performed confirm the presence or absence of UTI.
Assessment of patient quality of life. | week 0 (baseline), week 2 (after intervention), and week 4 （follow-up）
  Patient quality of life according to the EORTC QLQ-C30 scale. Higher scores on the functional subscales indicate better quality of life, whereas higher scores on the symptom subscales reflect more severe symptoms.

OTHER OUTCOMES:
Expectation evaluation | week 0 (baseline)
  Evaluation of Participants' Expectations. It can be understood as the proportion of participants who expect effective, ineffective, or unclear treatment outcomes.
Blinding evaluation | week 2 (after intervention)
  Blinding evaluation. It can be understood as the proportion of participants who are unaware of the intervention methods they have received.
Compliance evaluation | week 2 (after intervention), and week 4 （follow-up）
  Compliance evaluation. It can be understood as the proportion of participants who complete the study.
Safety evaluation | week 2 (after intervention), and week 4 （follow-up）
  Safety evaluation.The proportion of participants experiencing adverse events such as needle pain and subcutaneous hematoma.

IPD SHARING:
Plan to Share IPD: No